CLINICAL TRIAL: NCT01718275
Title: Non-operative Management of Early Appendicitis in Children
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Peter Minneci (Other)
Responsible Party: Sponsor-Investigator, Peter Minneci, Principal Investigator, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: IRB12-00406
Record Dates: First submitted 2012-10-29; First posted 2012-10-31 (Estimated); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Appendicitis
Keywords: Appendicitis; Pediatrics; Children; Non-operative
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Non-operative Group: Patients and caregivers who agree to receive non-operative management with antibiotics alone
- Surgery Group: Patients and caregivers who decide to undergo appendectomy that permit us to track their standard treatment course

SUMMARY:
The purpose of this study is to determine the feasibility of non-operative management of early appendicitis in children. We hypothesize that non-operative management of early appendicitis in children with antibiotics alone will be successful in 80% of children at 1 year follow-up.

DETAILED DESCRIPTION:
Non-operative management of appendicitis with antibiotics alone has recently emerged as a viable treatment alternative to appendectomy. There have been several clinical trials in adults which conclude that antibiotics alone are a safe initial treatment for appendicitis; none of these studies included children.

The primary objective of this study is to determine: conversion to surgery (failure of nonoperative management), 30 day, 6 month and 1 year recurrence rate of appendicitis in children treated with non-operative management. Recurrence is defined as need for appendectomy. The secondary objective is to compare adverse outcomes, length of stay, days to return to school, costs of care and quality of life measures between the study group and those that receive standard of care.We hypothesize that non-operative management of early appendicitis in children with antibiotics alone will be successful in 80% of children at 1 year follow-up.

This is a prospective, non-randomized single-site trial measuring the feasibility of treating children (7-17 years old) with early appendicitis with antibiotics only (non-operative management). There will be two cohorts; those who agree to receive non-operative management (Non-Operative Group) and those that permit us to track their standard treatment course (Surgery Group).

ELIGIBILITY:
Inclusion Criteria:

* Age : 7-17 years
* Ultrasound (US) or CT scan confirmed early appendicitis (US: hyperemia, <1.1 cm in diameter, compressible or non-compressible, no abscess, no fecalith, no phlegmon; CT: hyperemia, fat stranding, <1.1 cm in diameter, no abscess, no fecalith, no phlegmon)
* White blood cell count (WBC) < 15,000
* C reactive protein (CRP) <4 (if obtained)
* Focal abdominal pain </= 36 hours prior to receiving antibiotics

Exclusion Criteria:

* English is not the primary language of either the child or parent/guardian
* Other significant co-morbidities: cardiovascular disease, malignancy, pulmonary disease, diabetes, obesity (BMI ≥ 95th percentile for age and sex), severe developmental delay
* Positive urine pregnancy test
* Diffuse peritonitis
* Fecalith
* History of chronic intermittent abdominal pain
* WBC >/= 15
* CRP>/= 4 (if obtained)
* Pain > 36 hours prior to first antibiotic dose or any evidence on imaging studies concerning for evolving perforated appendicitis including abscess or phlegmon

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children treated a tertiary care Children's Hospital
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2014-02 (Actual); Study Completion 2023-08-22 (Estimated)

PRIMARY OUTCOMES:
Failure of Non-operative management | 1 year
  The primary endpoints are: conversion to surgery (failure of nonoperative management), 30-day, 6 month and one year recurrence rate.

SECONDARY OUTCOMES:
Adverse Outcomes | 1 year
  The secondary endpoints are: adverse outcomes, length of stay, days to return to school, costs of care and quality of life measures.

CONTACTS AND LOCATIONS:
Overall Officials: Peter C Minneci, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Minneci PC, Mahida JB, Lodwick DL, Sulkowski JP, Nacion KM, Cooper JN, Ambeba EJ, Moss RL, Deans KJ. Effectiveness of Patient Choice in Nonoperative vs Surgical Management of Pediatric Uncomplicated Acute Appendicitis. JAMA Surg. 2016 May 1;151(5):408-15. doi: 10.1001/jamasurg.2015.4534. PMID 26676711
- [Result] Minneci PC, Sulkowski JP, Nacion KM, Mahida JB, Cooper JN, Moss RL, Deans KJ. Feasibility of a nonoperative management strategy for uncomplicated acute appendicitis in children. J Am Coll Surg. 2014 Aug;219(2):272-9. doi: 10.1016/j.jamcollsurg.2014.02.031. Epub 2014 Apr 13. PMID 24951281